CLINICAL TRIAL: NCT06429137
Title: A Partially Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 3731579 Administered as Tablet to Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 3731579 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1519-0001; 2023-510318-25-00 (Registry Identifier: CTIS); U1111-1304-0523 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-05-21; First posted 2024-05-24 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BI 3731579 dose group 1 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 2 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 3 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 4 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 5 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 6 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 7 (Experimental)
  Interventions: Drug: BI 3731579
- BI 3731579 dose group 8 (Experimental)
  Interventions: Drug: BI 3731579
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo to BI 3731579

INTERVENTIONS:
Drug: BI 3731579 — BI 3731579
  Arms: BI 3731579 dose group 1; BI 3731579 dose group 2; BI 3731579 dose group 3; BI 3731579 dose group 4; BI 3731579 dose group 5; BI 3731579 dose group 6; BI 3731579 dose group 7; BI 3731579 dose group 8
Drug: Matching placebo to BI 3731579 — Matching placebo to BI 3731579
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 3731579 in healthy male subjects.

ELIGIBILITY:
Inclusion criteria

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 45 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion criteria

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 14 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 4 days
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com